CLINICAL TRIAL: NCT00399867
Title: Determination of the Efficacy and Feasibility of Simvastatin as Inhibitor of Cell Adhesion Mediated Drug Resistance in Patients With Refractory Multiple Myeloma - a Phase II Clinical Trial.
Brief Title: Simvastatin as Inhibitor of Cell Adhesion Mediated Drug Resistance in Patients With Refractory Multiple Myeloma.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SIMVA-272/04; Simva2005; 272/04
Record Dates: First submitted 2006-11-14; First posted 2006-11-15 (Estimated); Last update posted 2006-12-20 (Estimated); Status verified 2006-11

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma; refractory; cell adhesion mediated drug resistance
MeSH Terms: conditions — Multiple Myeloma | interventions — Simvastatin

INTERVENTIONS:
Drug: Simvastatin

SUMMARY:
In vitro statins, inhibitors of the HMG-CoA-reductase, have been shown to overcome cell adhesion mediated drug resistance at very low concentrations. The purpose of the study is to investigate the in vivo efficacy of simvastatin as inhibitor of cell adhesion mediated drug resistance. Patients refractory to ongoing chemotherapy will receive concomitantly simvastatin and response will be monitored by paraprotein levels

DETAILED DESCRIPTION:
Multiple Myeloma (MM) is an incurable haematological neoplasm that is characterized by homing, survival, and proliferation of malignant, antibody producing plasma cells in the bone marrow. All clinically relevant symptoms (cytopenia, hyperproteinemia and proteinuria with renal insufficiency, hypercalcemia, osteolysis) are due to the aggressive infiltration of the whole bone marrow by MM cells, while all other solid and lymphoid organs including the peripheral blood are normally spared. From these clinical observations and from many preclinical studies it is evident that adhesion of MM cells to the bone marrow cells characterizes the biology of this disease. Adhesion of MM cells leads to the secretion of stimulatory cytokines,upregulation of adhesion molecules, proliferation of MM cells, and drug resistance.

Statins, like simvastatin, inhibit the 3-hydroxy-3-methylglutaryl-coenzyme A (HMG-CoA) reductase, which catalyzes the conversion of HMG-CoA to mevalonate. Interestingly, in MM models statins induce apoptosis, inhibit proliferation, overcome primary and secondary drug resistance, and synergize with cytotoxic drugs. Oligonucleotide microarray analyses demonstrated that de novo and acquired drug resistance are associated with an increase of HMG-CoA reductase gene expression. We have shown before that adhesion of MM cells to bone marrow stromal cells mediates strong multidrug resistance and that this can be overcome by co-treatment with simvastatin in non-toxic concentrations. Interestingly, statin induced apoptosis in MM cells is not hampered by adhesion to bone marrow stromal cells.

Based upon these comprehensive preclinical findings clinical trials to investigate the in-vivo antimyeloma activity of statins are urgently needed. Our in vitro studies demonstrated that inhibition of cell adhesion mediated drug resistance by simvastatin is possible at low concentrations of about 1µM. We therefore suggested that cell adhesion mediated drug resistance can be treated with approved doses of simvastatin (80mg daily). Consequently we initiate a pilot phase II trial to investigate feasibility and clinical effects of simvastatin concomitantly with chemotherapy as preparation for a randomized trial.

As the primary goal is to prove the hypothesis that simvastatin can overcome drug resistance in vivo only patients not responding to chemotherapy will be included. Chemotherapy is defined as bortezomib and bendamustin, as both are effective and approved drugs in the therapy of relapsed myeloma. Further inclusion criteria are age over 18 years, proven MM (serum protein below 11g/dl, life expectancy > 3 months) and treatment indication with measurable paraprotein. In the case of no change (paraprotein increase less than 25% and paraprotein decline less than 50%) after two cycles of bortezomib (one cycle: 1.3 mg/m2 d1,4,8,11) or bendamustin (one cycle: 100 mg/m2 d1+2) the patients will receive two further cycles with concomitant simvastatin treatment (80 mg daily starting two days before chemotherapy and stopping two days after chemotherapy). Exclusion criteria are severe organ failure and risk factors for rhabdomyolysis (untreated hypothyroidism, active liver disease, terminal renal insufficiency, acute infectious disease, myopathy, heriditary myopathy in the family history, alcohol abuse, comedication with itraconazole, ketoconazole, erythromycin, clarithromycin, HIV protease inhibitors, nefazodone, cyclosporine, fibrates, niacin, amiodarone, verapamil).

ELIGIBILITY:
Inclusion Criteria:

* proven multiple myeloma,
* refractory to ongoing chemotherapy (bortezomib,
* bendamustin dexamethasone),
* measurable paraprotein,
* serum protein below 11 g/dl,
* age over 18 years,
* life expectancy greater 6 months,
* contraception in women,
* expected compliance,
* written consent

Exclusion Criteria:

* severe heart failure,
* not controlled hypertension or diabetes,
* risk factors for rhabdomyolysis,
* creatinin kinase below 30ml/min,
* active liver disease,
* myopathy,
* allergy to simvastatin,
* pregnancy,
* acute infectious disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2005-04; Study Completion 2007-04

PRIMARY OUTCOMES:
antimyeloma activity as measured by the paraprotein
toxicity of simvastatin in combination with chemotherapy

SECONDARY OUTCOMES:
duration of remission, event free survival, overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Bertold Emmerich, MD, PhD, Principal Investigator — Medizinische Klinik Innenstadt, University Munich

REFERENCES:
- [Background] Schmidmaier R, Baumann P, Simsek M, Dayyani F, Emmerich B, Meinhardt G. The HMG-CoA reductase inhibitor simvastatin overcomes cell adhesion-mediated drug resistance in multiple myeloma by geranylgeranylation of Rho protein and activation of Rho kinase. Blood. 2004 Sep 15;104(6):1825-32. doi: 10.1182/blood-2003-12-4218. Epub 2004 May 25. PMID 15161667